CLINICAL TRIAL: NCT04711070
Title: Understanding the Mechanisms of Critical Illness Myopathy by Use of a Novel Electrophysiological Method - Muscle Velocity Recovery Cycles (MVRCs)
Brief Title: Understanding the Mechanisms of Critical Illness Myopathy by Use of a Novel Electrophysiological Method - MVRCs
Status: Completed | Type: Observational
Sponsor: Sándor Beniczky (Other)
Collaborators: Danish Council for Independent Research (Other); University of Aarhus (Other); Søster og Verner Lipperts Fond (Unknown)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: MCIM
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Critical Illness Myopathy; Myopathy Critical Illness
Keywords: Critical Illness Myopathy; Muscle Velocity Recovery Cycles; Intensive Care Unit; Sepsis; Diagnosis; Pathophysiology
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with sepsis: Muscle velocity recovery cycles, electromyography, nerve conduction studies, direct musclestimulation, blood test
- Patients with chronic renal failure
- Healthy control

SUMMARY:
Critical illness myopathy (CIM) is a disabling condition that develops in critically ill patients. The syndrome is not only a cause of prolonged intensive care hospitalisation but also a main reason for delayed recovery. Critical illness myopathy presents as diffuse muscle weakness and failure to wean from mechanical ventilation.

The pathogenesis of CIM is unclear. The proposed mechanisms for critical illness myopathy include muscle membrane depolarization, circulating depolarizing factor, and an endotoxin that reduces muscle sodium channel availability at depolarized membrane potentials.

The electrophysiological diagnosis of CIM diagnosis is done by electromyography (EMG). In order to be able to detect changes in EMG, more than 2-3 weeks' time is required. Moreover the findings resemble other myopathies and are unspecific. EMG studies in paralysed muscles and sometimes unconscious patients is difficult or even impossible

Since the 1950s, it has been attempted to investigate the muscle cell membrane properties, but it has not been possible to develop a clinically applicable diagnostic method. The novel electrophysiological method MVRCs is a possible future diagnostic method. It's more sensitive to muscle cell membrane changes than existing methods and it is simple enough to use in multiple clinical settings.

The objective of this study is to investigate the utility of MVRCs in the early diagnosis of critical illness myopathy by investigating the muscle membrane properties in sepsis patients, who are in risk of developing CIM. In addition, this will contribute to a better understanding of the pathophysiology of critical illness myopathy.

The study will enrol 70 participants in total, divided in to 2 groups of 20 patients aged ≥18 years; 1) patients with sepsis at intensive care units and 2) patients with chronic renal failure and uremia, and 30 sex- and aged-matched healthy participants. All subjects are to undergo neurological examinations, electromyography, nerve conduction studies, direct muscle stimulation and MVRCs. Blood tests will be taken in all patients. Patients with sepsis will be examined every week in 3 weeks. The presence of probable CIM will be determined on the 4th examination. Healthy participants and patients with chronic renal failure will only be examined in 1 occasion.

The primary outcomes will be MVRCs parameters which will be compared between patients and healthy participants. Furthermore, MVRCs parameters will be correlated to blood sample results.

ELIGIBILITY:
Inclusion Criteria:

Patients: Fulfilled sepsis criteria of an increase in the Sequential (Sepsisrelated) Organ Failure Assessment (SOFA) score of 2 points or more.

Exclusion Criteria:

Patients and controls:

* Earlier peripheral nervous system disease
* History of malignancy, diabetes mellitus, alcoholism, medicine or other causes of polyneuropathy or myopathy
* Bleeding tendency or anticoagulation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients: Recruited from patients hospitalized in Intensive Care Units at the Department of Anaesthesiology and Intensive Care, Aarhus University Hospital.
  Healthy participants: Recruitment posters at Aarhus University, Aarhus University Hospital and at http://www.forsoegsperson.dk/.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2024-02-01 (Actual)

PRIMARY OUTCOMES:
Muscle relative refractory period (MRRP) | 12 weeks
  Measurement of changes in muscle membrane properties by MVRCs.
Early supernormality (ESN) | 12 weeks
  Measurement of changes in muscle membrane properties by MVRCs.

SECONDARY OUTCOMES:
Late supernormality (LSN) | 12 weeks
  Measurement of changes in muscle membrane properties by MVRCs.
Extra late supernormality (XLSN) | 12 weeks
  Measurement of changes in muscle membrane properties by MVRCs.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice H Tankisi, MD, PhD, Study Chair — Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Anaesthesiology and Intensive Care, Aarhus University Hospital, Aarhus C
  - Department of Clinical Neurophysiology, Aarhus University Hospital, Aarhus C